CLINICAL TRIAL: NCT06775405
Title: A Randomized, Double-blind, Placebo-controlled, Phase III Confirmatory Study to Evaluate the Efficacy, Safety, Tolerability, and Antiviral Activity of Repeated Oral Administration of AK0529 in Hospitalized Infants with Respiratory Syncytial Virus Infection
Brief Title: A Study to Confirm the Effectiveness and Safety of AK0529 in Treating RSV Infections in Hospitalized Infants
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Ark Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AK0529-2007
Record Dates: First submitted 2024-12-16; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Respiratory Synctial Virus Infections
MeSH Terms: interventions — ziresovir

STUDY DESIGN:
Intervention Model Description: This clinical study is a randomized placebo controlled parallel multi-center phase III trial.
Who Masked: Participant, Investigator
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active drug (Experimental): The participants will receive AK0529 of 10 mg, 20 mg or 40 mg based on body weight twice daily for 5 days from D1 to D5.
  Interventions: Drug: AK0529
- Placebo (Placebo Comparator): The participants will receive placebo of 10 mg, 20 mg or 40 mg based on body weight twice daily for 5 days from D1 to D5.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AK0529 — Active Substance: AK0529, Pharmaceutical Form: Enteric pellets, Route of Administration: Oral
  Arms: Active drug
Drug: Placebo — Active Substance: Placebo, Pharmaceutical Form: Enteric pellets, Route of Administration: Oral
  Arms: Placebo

SUMMARY:
Respiratory syncytial virus (RSV) is the most common respiratory infectious pathogen recognized worldwide that poses serious health risks to infants, and an important cause of hospitalization for severe respiratory infections in infants. Serious respiratory problems such as pneumonia caused by RSV are one of the leading causes of death from respiratory diseases in infants. AK0529 targets the Pre-F (fusion) protein on the surface of the viral envelope. Specifically, it prevents the virus from invading uninfected cells and inhibits the fusion between host cells by inhibiting the fusion of the F (fusion) proteins on the surface of the RSV envelope, thus providing the effects of anti-RSV infection. This is a randomized, double-blind, placebo-controlled, multicenter, phase III clinical study to evaluate the efficacy and safety of AK0529 in hospitalized infants aged 1 to 24 months with RSV infection. Considering the benefits of AK0529 in the population with RSV infection, hospitalized infants with moderate to severe RSV infection were selected as the target population for this study.

DETAILED DESCRIPTION:
This is a Phase III, randomized, double-blind, placebo-controlled, multicenter clinical study conducted among Chinese infants aged 1 to 24 months hospitalized with Respiratory Syncytial Virus (RSV) infection.

The study plans to enroll 180 infants aged 1 to 24 months with RSV infection. Eligible subjects will be randomized in a 1:1 ratio (AK0529: placebo). These subjects will receive the study drug twice daily for 5 consecutive days and the dose depends on subject's weight range.

Each subject in this study will undergo a visit schedule comprising a screening period of 36 hours before the first dose, a 5-day double-blinded treatment period, and a 9-day safety follow-up period after the last dose of treatment. The expected duration of participation for each subject will not exceed 17 days.

Infants successfully enrolled in this study will take the medication every 12 hours for 5 consecutive days, in total 10 doses. Investigators will regularly score the infants using the Wang bronchiolitis clinical score which is the primary endpoint. Additionally, nasopharyngeal aspirates samples will be collected from the infants for virological testing before the first dose on Days 1 to 5, on Day 6, and on Day 14.

Safety and tolerability assessments in this study will include evaluations of adverse events (AEs)/serious adverse events (SAEs), vital signs and blood oxygen saturation (SpO2) levels, physical examinations, clinical laboratory tests, and electrocardiogram (ECG) findings.

ELIGIBILITY:
Main Inclusion criteria:

1. Male or female subjects of any ethnicity with an age adjusted for any prematurity of ≥1 month and ≤24 months.
2. Diagnosis of RSV infection by any virological means, including a rapid diagnostic point-of-care testing, within 36 hours preceding initial dosing.
3. The onset of RSV infection symptoms should be ≤ 5 days prior to initial dosing.
4. Subject must weigh ≥ 2.5 kg and ≤ 20 kg at screening and be within the normal range for the subject's age, based on local child growth standards.
5. Subject must have a Wang bronchiolitis clinical score ≥ 5.

Main Exclusion criteria:

1. The subject has taken any restricted medications within 3 days prior to the date of screening or requires any restricted medications during treatment phase (including interferons, ribavirin, or proprietary Chinese medicines with antiviral effects) and has taken any inhaled or systemic glucocorticoids within 24 hours.
2. Subject is known to have co-infection with influenza virus, Mycoplasma, or other respiratory tract pathogens that require targeted clinical treatment .
3. Subject is known to have bacterial pneumonia.
4. Subject with clinical evidence of hepatic decompensation (e.g., liver disease with coagulation abnormalities or encephalopathy).
5. Subject with inborn symptoms of metabolic abnormalities (e.g., mitochondrial diseases, carbohydrate metabolism abnormalities, glycogen accumulation diseases).
6. Subject with chronic or persistent feeding difficulties.
7. The parent or guardian of the subject is an employee of the study investigator or the study facility (such person will be directly involved in the study or any other study administered by the study facility investigator), or a family member of the study investigator or his/her staff.
8. Subject who have participated in clinical trials of other drugs or devices in the 30 days prior to screening.
9. Subject with any other reason that the investigator deems unsuitable for participation in the study.

Ages: 1 Month to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2024-02-29 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the Wang bronchiolitis clinical score | Day 3 (48 hours)
  The Wang bronchiolitis clinical score will be used to evaluate respiratory rate, wheezing, respiratory muscle retraction and "general condition" (sleep, feeding, and general status) in subjects with symptoms of bronchiolitis. Each item of the scale is divided into 4 levels according to the severity of symptoms, with 0 point indicating normal and 3 points the highest severity, 12 points in total.

SECONDARY OUTCOMES:
Change from baseline in the Wang bronchiolitis clinical score in subjects younger than 6 months. | Day 3 (48 hours)
  The Wang bronchiolitis clinical score will be used to evaluate respiratory rate, wheezing, respiratory muscle retraction and "general condition" (sleep, feeding, and general status) in subjects with symptoms of bronchiolitis. Each item of the scale is divided into 4 levels according to the severity of symptoms, with 0 point indicating normal and 3 points the highest severity, 12 points in total.
Time from first treatment to sustained remission of symptoms during the treatment period. | Study period (up to 14 days)
  The sustained remission is defined as achieving a total Wang bronchiolitis clinical score of 0 or 1 for 48 consecutive hours without support of oxygen therapy.
Change in RSV VL (viral load) from baseline at each visit. | Day 2, Day 3, Day 4, Day 5, Day 6, Day 14
  The viral load of subjects' nasopharyngeal samples will be measured by quantitative reverse transcription polymerase chain reaction (qRT-PCR).
Proportion of subjects with RSV VL below the lower limit of quantitation (LLOQ) at each visit. | Day 2, Day 3, Day 4, Day 5, Day 6, Day 14
  The viral load of subjects' nasopharyngeal samples will be measured by quantitative reverse transcription polymerase chain reaction (qRT-PCR).
Time from first treatment to mild disease for subjects, defined as achieving a Wang bronchiolitis clinical score ≤ 3 without the need for supplemental oxygen. | Study period (up to 14 days)
Change in sub-scores of the Wang bronchiolitis clinical score from baseline at each visit. | Day 2, Day 3, Day 4, Day 5, Day 6, Day 14
  The Wang bronchiolitis clinical score will be used to evaluate respiratory rate, wheezing, respiratory muscle retraction and "general condition" (sleep, feeding, and general status) in subjects with symptoms of bronchiolitis. Each item of the scale is divided into 4 levels according to the severity of symptoms, with 0 point indicating normal and 3 points the highest severity, 12 points in total.
Time from initial dosing to resolution of symptoms based on sub-scores of the Wang bronchiolitis clinical score. | Study period (up to 14 days)
  The resolution is defined as achieving the following sub-scores without the need for supplemental oxygen:
  * Respiratory rate = 0 or 1
  * Wheezing = 0 or 1
  * Respiratory muscle retraction = 0 or 1
  * General condition = 0 Note: The above indicators are only for subjects with a baseline sub-score greater than 0 for the respective sub-scores.
Safety endpoints | Study period (up to 14 days)
  The safety assessment includes the following events, tests, indicators occurring during the study process:
  * Incidence rate and severity of Adverse Events (AEs), Serious Adverse Events (SAEs), and withdrawal from the study due to AEs;
  * Laboratory tests;
  * Electrocardiogram (ECG);
  * Physical examination and vital signs.
Pharmacokinetic endpoints | Study period (up to 14 days)
  Include but not limit to steady state AUC, Cmax and Ctrough.

CONTACTS AND LOCATIONS:
Locations (17):
- China (17):
  - Beijing Children's Hospital, Capital Medical University, Beijing
  - First Hospital of Jilin University, Changchun
  - Hunan Provincial People's Hospital, Changsha
  - West China Second University Hospital, Sichuan University, Chengdu
  - Children's Hospital, Zhejiang University School of Medicine, Hangzhou
  - Sanya Central Hospital, Hainan Third People's Hospital, Sanya
  - Shanghai Children's Hospital, Shanghai Jiao Tong University, Shanghai
  - Shanghai Children's Medical Center, Shanghai Jiao Tong University School of Medicine, Shanghai
  - Shengjing Hospital of China Medical University, Shenyang
  - Tianjin Children's Hospital（Longyan）, Tianjin
  - Tianjin Children's Hospital（Machang）, Tianjin
  - Second Affiliated Hospital and Yuying Children's Hospital of Wenzhou Medical University, Wenzhou
  - Wuhan Children's Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - Wuxi Children's Hospital, Wuxi
  - First Affiliated Hospital of Xiamen University, Xiamen
  - Women and Children's Hospital, and the School of Medicine, Xiamen University, Xiamen
  - Zhongshan Women and Children's Hospital-Zhongshan Boai Hospital, Zhongshan

IPD SHARING:
Plan to Share IPD: No